CLINICAL TRIAL: NCT01317485
Title: Laparoscopic Peritoneal Lavage or Resection for Generalised Peritonitis for Perforated Diverticulitis: a Nationwide Multicenter Randomised Trial
Brief Title: Laparoscopic Peritoneal Lavage or Resection for Generalised Peritonitis for Perforated Diverticulitis
Acronym: Ladies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Prof. dr. W.A. Bemelman / Prof. dr. J.F. Lange, Academic Medical Centre Amsterdam / Erasmus Medical Centre Rotterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTR2037
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Perforated Diverticulitis
Keywords: diverticulitis; perforation; sigmoidectomy; sigmoid resection; lavage; laparoscopic; wash-out; rinsing; hartmann; end-colostomy; primary anastomosis
MeSH Terms: conditions — Diverticulitis | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Purulent peritonitis (Experimental): Patients with purulent peritonitis are randomised at a 2:1:1 ratio between
  1. Laparoscopic lavage and drainage
  2. Sigmoidectomy with primary anastomosis
  3. Sigmoidectomy with end-colostomy
  Interventions: Procedure: Laparoscopic lavage and drainage; Procedure: Sigmoidectomy with primary anastomosis; Procedure: Sigmoidectomy with end-colostomy
- Fecal peritonitis or overt perforation (Experimental): Patients with fecal peritonitis or an overt perforation are randomised between
  1. Sigmoidectomy with primary anastomosis
  2. Sigmoidectomy with end-colostomy
  Interventions: Procedure: Sigmoidectomy with primary anastomosis; Procedure: Sigmoidectomy with end-colostomy

INTERVENTIONS:
Procedure: Laparoscopic lavage and drainage — [CLOSED] The abdominal cavity is irrigated with six litres of warm saline in all four quadrants. At the end of the procedure a Douglas drain is inserted via the right lateral port.
  ***This part of the study was closed in 2013 on advice of the data and safety monitoring board due to safety issues
  Arms: Purulent peritonitis
Procedure: Sigmoidectomy with primary anastomosis — [OPEN] Sigmoidectomy is done according to the guidelines of the American Society of Colon and Rectal Surgeons. The distal transsection margin has to be on the proximal rectum, the proximal margin is determined by the absence of wall thickening due to diverticulitis. The type of anastomosis is done according to the preference of the operating surgeon. A loop ileostomy can be fashioned in order to ensure faecal deviation to the discretion of the surgeon.
  Other Names: Sigmoid resection
Procedure: Sigmoidectomy with end-colostomy — [OPEN] This is a two-stage procedure with the intention to close the colostomy in a second stage. During the primary surgery, only the perforated diseased part must be resected. There is no need of having the distal transsection line on the proximal rectum.
  Other Names: Hartmann procedure

SUMMARY:
The first objective (LOLA) of this integrated trial is to determine whether laparoscopic lavage leads to better clinical outcomes compared to sigmoidectomy in patients with perforated diverticulitis with purulent peritonitis in terms of mortality and major morbidity. The second objective (DIVA) is to determine whether sigmoidectomy with anastomosis or sigmoidectomy with end-colostomy is the superior approach in patients with perforated diverticulitis with either purulent or faecal peritonitis in terms of stoma free survival. The study is designed as a multicenter and randomised trial.

DETAILED DESCRIPTION:
Patients diagnosed as having perforated diverticulitis with free air on plain abdominal X-ray or CT scan fulfilling the in- and exclusion criteria are randomised during laparoscopy via a central computer. In case of purulent diverticulitis patients are randomised to three arms: (a) laparoscopic lavage, (b) sigmoidectomy with colostomy or (c) sigmoidectomy with anastomosis in ratio of 2:1:1. In case of faecal peritonitis or an overt perforation of the sigmoid, the patient will be randomised 1:1 to sigmoidectomy with colostomy or sigmoidectomy with primary anastomosis.

The first primary outcome parameter consists of a combined endpoint consisting of mortality and major morbidity (LOLA). The second primary endpoint consists of stoma-free survival one year after initial surgery (DIVA). Secondary endpoints are number of days alive and outside the hospital, health related quality of life, health care utilisation and associated costs. A sample size of 132:66:66 patients per treatment arm will be able to detect a difference in the combined endpoint of serious complications and mortality from 25% in the two sigmoidectomy groups compared to 10% in the lavage group (two-side alpha of 5% and a power of 90%. In the DIVA analysis 2x132 patients are needed to significantly demonstrate a difference of 30% in stoma-free survival between both treatment arms (log rank test two-sided alpha of 5% and power of 90%) in favour of the patients with primary anastomosis. More than 35 hospitals will participate in this study with an estimated total inclusion of 100 patients per year. Patients will be followed for one year.

The study will be executed in concordance with the protocol, the Good Clinical Practice guidelines and regulatory requirements.

After closure of the LOLA-arm due to safety concerns for laparoscopic lavage, the protocol and sample size has for the DIVA-arm been adjusted to 118 patients per study arm (faecal or purulent peritonitis).

ELIGIBILITY:
Inclusion Criteria:

patients suspected of diverticulitis

* age in between 18 and 85 years old
* with written informed consent
* with free air on plain abdominal or thoracic X-ray or CT-scan OR with peritonitis and diffuse gas or fluid on CT-scan

Exclusion Criteria:

* dementia
* prior sigmoidectomy
* steroid treatment > 20 mg daily
* prior pelvic irradiation
* preoperative shock: requirement of inotropics due to circulatory insufficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Estimated)
Dates: Start 2010-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Mortality and major morbidity (combined) | One-year
  The primary outcome in the lavage vs. resectional intervention comparison (LOLA), will be poor clinical outcome, defined as a combined endpoint consisting of mortality and major morbidity one year after initial surgery. Major morbidity includes any of the following events or conditions: reintervention, wound dehiscence, incisional hernia, abscess needing percutaneous drainage, urosepsis, myocardial infarction, renal failure and respiratory insufficiency.
Stoma-free survival | One year
  Stoma-free survival one year after initial surgery, is the primary outcome for the comparison of the resectional strategies (DIVA).

SECONDARY OUTCOMES:
Operating time | - (day 1)
Hospital stay | - (day one until discharge from hospital)
Number of days alive and outside the hospital | One year
Incisional hernia | One year
Reinterventions | One year
  All reinterventions within a one year time frame, including percutaneous abscess drainage.
Health related quality of life | One year
  SF-36, EQ-5D, GIQLI measured at 2, 4, 13 and 26 weeks after primary surgery.
Health care utilisation and associated costs | One year
  SF-HLQ measured at 4, 13, 26, 39 and 52 weeks after primary surgery

CONTACTS AND LOCATIONS:
Overall Officials: J.F. Lange, Professor, Principal Investigator — Erasmus Medical Centre, Rotterdam; W.A. Bemelman, Professor, Principal Investigator — Academic Medical Centre, Amsterdam
Locations (41):
- Belgium (2):
  - University Clinic St. Luc, Brussels
  - University Hospital Leuven, Leuven
- Netherlands (39):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Flevo Hospital, Almere Stad
  - Rijnland Hospital, Alphen Aan de Rijn and Leiderdorp
  - Meander Medical Centre, Amersfoort
  - Academic Medical Centre, Amsterdam
  - Free University Medical Centre, Amsterdam
  - Onze Lieve Vrouwe Hospital, Amsterdam
  - Slotervaart Hospital, Amsterdam
  - St. Lucas Andreas Hospital, Amsterdam
  - Alysis Medical Centre, Arnhem
  - Rode Kruis Hospital, Beverwijk
  - Amphia Hospital, Breda
  - IJsselland Hospital, Capelle aan den IJssel
  - Reinier de Graaf Hospital, Delft
  - Deventer Hospital, Deventer
  - Albert Schweitzer Hospital, Dordrecht and Zwijndrecht
  - Gelderse Vallei Hospital, Ede
  - Catharina Hospital, Eindhoven
  - Medical Spectrum Twente, Enschede
  - Groene Hart Hospital, Gouda
  - Kennemer Hospital, Haarlem
  - Atrium Medical Centre, Heerlen and Brunssum
  - Tergooi Hospitals, Hilversum and Blaricum
  - Spaarne Hospital, Hoofddorp
  - Westfries Hospital, Hoorn
  - Leiden University Medical Centre, Leiden
  - Maastricht University Medical Centre, Maastricht
  - St. Antonius Hospital, Nieuwegein
  - Erasmus Medical Centre, Rotterdam
  - Ikazia Hospital, Rotterdam
  - Maasstad Hospital, Rotterdam
  - St. Franciscus Hospital, Rotterdam
  - Orbis Medical Centre, Sittard
  - Haga Hospital, The Hague
  - Twee Steden Hospital, Tilburg and Waalwijk
  - University Medical Centre Utrecht, Utrecht
  - Máxima Medical Centre, Veldhoven
  - Zaans Medical Centre, Zaandam
  - Isala Hospitals, Zwolle

REFERENCES:
- [Background] Toorenvliet BR, Swank H, Schoones JW, Hamming JF, Bemelman WA. Laparoscopic peritoneal lavage for perforated colonic diverticulitis: a systematic review. Colorectal Dis. 2010 Sep;12(9):862-7. doi: 10.1111/j.1463-1318.2009.02052.x. Epub 2009 Sep 26. PMID 19788490
- [Background] Salem L, Flum DR. Primary anastomosis or Hartmann's procedure for patients with diverticular peritonitis? A systematic review. Dis Colon Rectum. 2004 Nov;47(11):1953-64. doi: 10.1007/s10350-004-0701-1. PMID 15622591
- [Background] Constantinides VA, Tekkis PP, Athanasiou T, Aziz O, Purkayastha S, Remzi FH, Fazio VW, Aydin N, Darzi A, Senapati A. Primary resection with anastomosis vs. Hartmann's procedure in nonelective surgery for acute colonic diverticulitis: a systematic review. Dis Colon Rectum. 2006 Jul;49(7):966-81. doi: 10.1007/s10350-006-0547-9. PMID 16752192
- [Derived] Hoek VT, Edomskis PP, Stark PW, Lambrichts DPV, Draaisma WA, Consten ECJ, Lange JF, Bemelman WA; LADIES trial collaborators. Laparoscopic peritoneal lavage versus sigmoidectomy for perforated diverticulitis with purulent peritonitis: three-year follow-up of the randomised LOLA trial. Surg Endosc. 2022 Oct;36(10):7764-7774. doi: 10.1007/s00464-022-09326-3. Epub 2022 May 23. PMID 35606544
- [Derived] Lambrichts DPV, Vennix S, Musters GD, Mulder IM, Swank HA, Hoofwijk AGM, Belgers EHJ, Stockmann HBAC, Eijsbouts QAJ, Gerhards MF, van Wagensveld BA, van Geloven AAW, Crolla RMPH, Nienhuijs SW, Govaert MJPM, di Saverio S, D'Hoore AJL, Consten ECJ, van Grevenstein WMU, Pierik REGJM, Kruyt PM, van der Hoeven JAB, Steup WH, Catena F, Konsten JLM, Vermeulen J, van Dieren S, Bemelman WA, Lange JF; LADIES trial collaborators. Hartmann's procedure versus sigmoidectomy with primary anastomosis for perforated diverticulitis with purulent or faecal peritonitis (LADIES): a multicentre, parallel-group, randomised, open-label, superiority trial. Lancet Gastroenterol Hepatol. 2019 Aug;4(8):599-610. doi: 10.1016/S2468-1253(19)30174-8. Epub 2019 Jun 6. PMID 31178342
- [Derived] Vennix S, Musters GD, Mulder IM, Swank HA, Consten EC, Belgers EH, van Geloven AA, Gerhards MF, Govaert MJ, van Grevenstein WM, Hoofwijk AG, Kruyt PM, Nienhuijs SW, Boermeester MA, Vermeulen J, van Dieren S, Lange JF, Bemelman WA; Ladies trial colloborators. Laparoscopic peritoneal lavage or sigmoidectomy for perforated diverticulitis with purulent peritonitis: a multicentre, parallel-group, randomised, open-label trial. Lancet. 2015 Sep 26;386(10000):1269-1277. doi: 10.1016/S0140-6736(15)61168-0. Epub 2015 Jul 22. PMID 26209030
- See also: Related Info — http://www.diverticulitis.nl